CLINICAL TRIAL: NCT02191657
Title: A Double Blind, Placebo-controlled, Dose-escalating, Multiple Dose Study, Investigating the Safety, Antiretroviral Activity, Tolerability and Pharmacokinetic Profile of Deferiprone When Administered in Healthy Volunteers and Asymptomatic HIV Infected Subjects
Brief Title: Antiretroviral Activity and Pharmacokinetics of Deferiprone in Healthy Volunteers and Asymptomatic HIV-infected Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ApoPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: LA26-106
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2007-11

CONDITIONS: HIV Infection
Keywords: HIV; deferiprone; iron chelation
MeSH Terms: conditions — HIV Infections | interventions — Deferiprone; Long Interspersed Nucleotide Elements

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): Subjects in this arm were asymptomatic HIV-infected individuals who received a dose of 33 mg/kg deferiprone three times a day for a total daily dosage of 99 mg/kg
  Interventions: Drug: Deferiprone
- Cohort 2 (Experimental): Subjects in this arm were healthy volunteers who received a dose of 50 mg/kg deferiprone three times a day for a total daily dosage of 150 mg/kg
  Interventions: Drug: Deferiprone
- Cohort 3 (Experimental): Subjects in this arm were asymptomatic HIV-infected individuals who received a dose of 50 mg/kg deferiprone three times a day for a total daily dosage of 150 mg/kg.
  Interventions: Drug: Deferiprone

INTERVENTIONS:
Drug: Deferiprone — Oral iron chelator
  Other Names: Ferriprox; L1

SUMMARY:
The purpose of this study was to examine the safety, efficacy, and pharmacokinetics of different dosages of deferiprone in subjects with or without HIV infection.

DETAILED DESCRIPTION:
Three cohorts were enrolled: two of individuals who were asymptomatically infected with HIV and one of healthy volunteers. Dosages were as follows:

* Cohort 1 (asymptomatic HIV infected subjects): 33 mg/kg deferiprone three times daily for a total of 99 mg/kg/day
* Cohort 2 (healthy volunteers): 50 mg/kg deferiprone three times daily for a total of 150 mg/kg/day
* Cohort 3 (asymptomatic HIV infected subjects): 50 mg/kg deferiprone three times daily for a total of 150 mg/kg/day

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥18 years and ≤ 60 years.
* Absolute neutrophil count (ANC) of >1000/mm3 for African black population and ≥ 1600/mm3 for all other races.
* For Cohort 2: HIV-negative
* For Cohorts 1 and 3: HIV-1 positive; CD4 count of at least 300/mm3; HIV-1 RNA copies (viral load) >10 000 copies/mL serum; and current physical health stable and not requiring antiretroviral treatment
* For Cohorts 1 and 3: Chest x-ray showing absence of active infectious diseases (such as tuberculosis, viral or atypical bacteria or parasitic infection).

Exclusion Criteria:

* Presence of any severe concomitant disease.
* History of or current, recurrent or recent (4 weeks) febrile disease.
* History of opportunistic infections, neoplasm or AIDS-defining conditions.
* Inability to discontinue any medication from screening onwards, or for at least 2 weeks before the first admission; in particular any antiviral or therapy with immunosuppressive activity.
* Significant liver impairment: aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≥ 2.5 times the upper normal limit.
* Significant kidney impairment: serum creatinine ≥ two times the upper normal limit.
* Any concomitant disorder or resultant therapy likely to have interfered with subject compliance or with study procedures.
* Known hypersensitivity to any of the test materials or related compounds.
* Positive test for Hepatitis B and/or C antibodies.
* A history of multiple and/or severe allergies to drugs or foods or a history of anaphylactic reactions.
* History of seizures or epilepsy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2006-11; Primary Completion 2008-05 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events following repeated oral doses of deferiprone in asymptomatic HIV-infected subjects and healthy volunteers | 9 weeks (from receipt of first dose until 8 weeks after the last dose)
  Collection of adverse events, including abnormal findings in physical examination, vital signs, 12-lead ECG, 24-hour Holter ECG, and laboratory variables (hematology, clinical chemistry, and urinalysis)
Measurement of viral load following repeated oral doses of deferiprone in asymptomatic HIV-infected subjects and healthy volunteers | 9 weeks (pre-dose until 8 weeks after last dose)
  Measurement of HIV RNA load for the assessment of antiretroviral activity
Cluster of differentiation 4 (CD4) count and p24 antigen status following repeated oral doses of deferiprone in asymptomatic HIV-infected subjects and healthy volunteers | 1 week (pre-dose to day of last dose)
  Measurement of CD4 count and p24 antigen status for assessment of antiviral activity

SECONDARY OUTCOMES:
Cmax of deferiprone and deferiprone 3-O-glucuronide | 24-hour interval
  Determination of Cmax following a dose of deferiprone in asymptomatic HIV-infected subjects and healthy volunteers
Tmax of deferiprone and deferiprone 3-O-glucuronide | 24-hour interval
  Determination of Tmax of deferiprone and its metabolite following a dose of deferiprone in asymptomatic HIV-infected subjects and healthy volunteers
Area under the curve (AUC) 0-infinity of deferiprone and deferiprone 3-O-glucuronide | 24-hour interval
  Determination of AUC 0-infinity of deferiprone and its metabolite following a dose of deferiprone in asymptomatic HIV-infected subjects and healthy volunteers
T1/2 of deferiprone and deferiprone 3-O-glucuronide | 24-hour interval
  Determination of T1/2 of deferiprone and its metabolite following a dose of deferiprone in asymptomatic HIV-infected subjects and healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Dewald Steyn, MD, Principal Investigator — University of the Free State, South Africa
Locations (1):
- PAREXEL International, Bloemfontein, South Africa

REFERENCES:
- [Derived] Saxena D, Spino M, Tricta F, Connelly J, Cracchiolo BM, Hanauske AR, D'Alliessi Gandolfi D, Mathews MB, Karn J, Holland B, Park MH, Pe'ery T, Palumbo PE, Hanauske-Abel HM. Drug-Based Lead Discovery: The Novel Ablative Antiretroviral Profile of Deferiprone in HIV-1-Infected Cells and in HIV-Infected Treatment-Naive Subjects of a Double-Blind, Placebo-Controlled, Randomized Exploratory Trial. PLoS One. 2016 May 18;11(5):e0154842. doi: 10.1371/journal.pone.0154842. eCollection 2016. PMID 27191165